CLINICAL TRIAL: NCT05468827
Title: ICG Fluorescence Guided Lymph Node Mapping for Determination of Bowel Resection Margins in Colon Cancer
Acronym: ISCAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ISC-1
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Colon Cancer
Keywords: colon cancer; lymphatic mapping; indocyanine green
MeSH Terms: conditions — Colonic Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: all study participants are allocated to intraoperative ICG mapping of locoregional lymphatic collector
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interventional (Experimental): lymphatic mapping by indocyanine green
  Interventions: Procedure: lymphatic mapping with indocyanine green

INTERVENTIONS:
Procedure: lymphatic mapping with indocyanine green — subserosal injection of indocyanine green near the primary tumour with subsequent assessment of the dye spread along lymphatics

SUMMARY:
The study is aimed at investigating feasibility of defining colon resection margins for colon cancer with ICG by comparing lymphatic distribution of subserosally injected dye with actual spread of lymphatic metastases reported by pathologists after specimen examination

DETAILED DESCRIPTION:
In this study 2.5 mg/ml indocyanine green solution is injected subserosally into colonic wall near the tumour in 4 points (1 ml each). The fluorescence is assessed before specimen removal (at least 30 min after injection) and its mesenteric distribution is marked by surgeon on the specimen. Proximal and distal colonic resection margins are chosen to be at least 10 cm long and to include the whole area of fluorescence. After removal, lymphatic node groups according JSCCR are also marked on fresh specimen. During pathological examination each lymph node is assessed not only for presence of metastases but also for its exact location in relation to margins of indocyanine distribution.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed adenocarcinoma of colon (caecum, ascending colon, hepatic flexure, transverse colon, splenic flexure, descending colon, sigmoid)
2. TNM T1-4a N0-2 M0-1
3. Clinical indications to colonic resection
4. ECOG - 0-2
5. Signed informed consent.

Exclusion Criteria:

1. Medical or psychiatric reasons interfering with patient's decision to participate in the study.
2. Pregnancy or breastfeeding.
3. Medical conditions contraindicating surgical procedure.
4. Acute bowel obstruction, bleeding or perforation.
5. Hypersensitivity to indocyanine green, sodium iodide or iodine
6. Hyperthyroidism or autonomic thyroid adenomas
7. Kidney failure of any aetiology
8. Hepatic failure of any aetiology
9. Poorly tolerated indocyanine injection in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
proportion of pN+ patients in which affected lymph nodes are detected only within margins of ICG distribution | 30 days
  number of patients with affected lymph nodes located within ICG distribution margins divided by the number of all patients with pN+

SECONDARY OUTCOMES:
incidence of adverse events related to ICG lymphatic mapping | 30 days
  proportion of patients facing adverse events related to ICG lymphatic mapping procedure
feasibility of ICG lymphatic mapping for colon cancer | duration of surgical procedure
  proportion of ICG spillage affecting interpretation
incidence of lymph node metastases outside conventional resection margins (10 cm) | 30 days
  proportion of patients with aberrant lymphatics leading to affected lymph nodes
colon cancer lymphatic spread pattern | 30 days
  descriptive data on incidence of D1, D2 and D3 lymphatic collector metastases and frequences of D1 collector metastases depending on distance from primary tumour
feasibility of ICG mapping for colon flexure tumours | duration of surgical procedure
  proportion of operations for colon flexure tumours which extent is effected by ICG lymphatic mapping

CONTACTS AND LOCATIONS:
Overall Officials: Aleksey Karachun, PhD, Study Director — N.N. Petrov National Medicine Research Center of oncology
Locations (1):
- N.N. Petrov National Medical Research Center of Oncology, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No